CLINICAL TRIAL: NCT02356744
Title: Comparison of Maternal and Neonatal Outcome Before and After 1 Year of Bariatric Surgery
Brief Title: Maternal and Neonatal Outcome in Pregnant Women Before and After 1 Year Since Bariatric Operation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 126
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy, Complications
Keywords: Maternal outcome; Fetal outcome; bariatric surgery; Third Trimester
MeSH Terms: conditions — Pregnancy Complications | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- surgery done less than 1 year: Pregnant women who had bariatric surgery done within the last year before pregnancy. Ultrasound fetal monitoring,biophysical profile assessment and maternal follow up investigations and blood pressure monitoring through all pregnancy
  Interventions: Other: Ultrasound
- surgery done more than 1 year: Pregnant women who had bariatric surgery done more than 1 year before pregnancy. Ultrasound fetal monitoring,biophysical profile assessment and maternal follow up investigations and blood pressure monitoring through all pregnancy
  Interventions: Other: Ultrasound

INTERVENTIONS:
Other: Ultrasound — Ultrasound assessment of fetal growth, anomalies , liqour and placenta

SUMMARY:
Ultrasound follow up for 9 months pregnancy in women underwent baraitric surgery before and after 1 year of surgery.

DETAILED DESCRIPTION:
Ultrasound follow up for 9 months pregnancy in women who had laparoscopic adjustable gastric banding done within last 1 year or earlier.

ELIGIBILITY:
Inclusion Criteria:

* 1.Pregnant women in third trimester 2.after laparoscopic adjustable gastric banding done within last 1 year or earlier

Exclusion Criteria:

* medical disorders affecting pregnancy as diabetes, hypertension, SLE

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women in third trimester after laparoscopic adjustable gastric banding done within last 1 year or earlier
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02-02 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
maternal outcome | though 9 months of pregnancy and 6 weeks postpartum
  development of pregnancy complications as preeclampsia or gestational diabetes or postpartum complications as postpartum hemorrhage or puerperal sepsis

SECONDARY OUTCOMES:
Neonatal outcome | 2 weeks after birth
  Apgar score, neonatal ICU admission
Route of delivery | time of delivery
  vaginal delivery or cesarean section and if cesarean its indications

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt